CLINICAL TRIAL: NCT01096641
Title: An Explorative Study on Physiological and Neurophysiological Determinants of Fatigue in Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FICS 20084002
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Postcancer Fatigue
Keywords: Fatigued disease-free Cancer Patients; cancer treatment finished > one year and < ten years ago

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fatigued patients: Immediate start CBT (Other): After the baseline assessment the fatigued patients will be randomized to start immediately with Cognitive Behaviour Therapy, especially designed for fatigued cancer patients. At the end of the therapy, after 6 months, a second assessment will take place.This assessment will include the same measurements as at baseline.
  Interventions: Behavioral: immediate CBT
- fatigues patients: delayed CBT (after 6 months) (Other): The fatigued patients on the waiting list will start with CBT after 6 months
  Interventions: Behavioral: Delayed CBT
- non-fatiqued controls (No Intervention): Non-fatigued control group. This group is not included in the randomization.

INTERVENTIONS:
Behavioral: immediate CBT — After the baseline assessment the fatigued patients will be randomized to start immediately with Cognitive Behaviour Therapy, especially designed for fatigued cancer patients
  Arms: Fatigued patients: Immediate start CBT
Behavioral: Delayed CBT — After the baseline assessment the fatigued patients will be randomized: this group is to be placed on a waiting list. After 6 months, a second assessment will take place in the group of fatigued patients who received CBT immediately after randomization. This assessment will include the same measurements as at baseline. The fatigued patients on the waiting list will then start with CBT.
  Arms: fatigues patients: delayed CBT (after 6 months)

SUMMARY:
Postcancer fatigue is a severe and invalidating problem, impairing quality of life. About 20 to 40% of the patients remain fatigued, at least one year after successful cancer treatment. Fortunately, there is an effective treatment for postcancer fatigue; cognitive behavior therapy. However, no cause for postcancer fatigue has been identified yet. The aim of the study is to identify factors that (partly) cause postcancer fatigue to improve the theoretical understanding of fatigue and to improve the diagnostics of fatigue, predict therapy outcome, and facilitate other treatment options.

In this study, disease-free fatigued cancer patients, who finished treatment for cancer at least one year and maximally ten years ago, will be approached for this study. They will be compared to non-fatigued patients.

First, a baseline assessment will take place. Magnetic resonance imaging of the brains will be performed to assess brain volume and magnetic resonance spectroscopy will be performed to measure the concentrations of specific substances in the brains. Changes in the volume of parts of the brains have been observed in (non-cancer) patients with the chronic fatigue syndrome (CFS), in comparison with healthy controls. In addition, abnormal concentrations of specific substances have been observed in patients with CFS compared to healthy controls. To assess muscle fatigue, a two-minute endurance test of the upper arm will be administered at maximal voluntary contraction. Next to differences in the brains, CFS patients showed (central) muscle fatigue. A maximal exercise test on a bicycle will be performed to assess physical fitness. Physical activity in fatigued cancer survivors is decreased, compared to healthy controls. It is not known whether physical deconditioning originated during the cancer treatment is the reason why these patients are still less active. In addition, patients and controls will wear an actometer for two weeks to register baseline daily physical activity and for an additional 5 days after the maximal exercise test, to assess the effect of exercise on the daily physical activity. Finally, patients and controls will complete standardized questionnaires and will perform neurological/psychological tests, like a reaction time test and a short time memory task, at baseline.

The results of the non-fatigued and the fatigued patients will be compared at baseline. For the non-fatigued participants, the study will be finished after the baseline measurements. The fatigued participants will start with cognitive behavior therapy immediately after the baseline measurements or after 6 months, depending on the randomization.

At the end of the therapy, after six months, or after 6 months of waiting for cognitive behavior therapy, a second assessment will take place, comparable to the baseline measurements. These results will be compared with the baseline situation to analyze the effect of cognitive behavior therapy on the (possible) causes of postcancer fatigue.

DETAILED DESCRIPTION:
Fatigue after curative treatment for cancer is a severe and invalidating problem. 20-40% of disease-free cancer patients mention fatigue as a frequent complaint, impairing quality of life. In search for (neuro)physiological factors determining fatigue, our centre has recently demonstrated the presence of morphological differences in the brains of non-cancer patients with the chronic fatigue syndrome (CFS) compared with healthy volunteers. Both in patients with CFS and in fatigued patients with neuromuscular diseases we showed that fatigue has a central neurophysiological component (so-called central activation failure). Others have shown that chronic fatigue is associated with altered brain metabolism. Studies with proton MR spectroscopy (1H MRS) have demonstrated a higher choline to creatine ratio in the brains of chronically fatigued patients. This suggests increased cell membrane turnover. Also reduced levels of N-acetylaspartate-creatine ratio (NAA/Cr) in the right hippocampus have been observed in these patients, which suggests a decrease in functional axons. Finally, elevated ventricular lactate was observed, which suggests changes in brain glucose metabolism. Actigraphy has shown that actual physical activity in fatigued cancer survivors is decreased compared to healthy controls. It is not known whether physical deconditioning originated during the actual cancer treatment is the reason why these patients are still less active. Until now no other (neuro)physiological factors have been identified explaining fatigue in cancer survivors. Recently we have shown that Cognitive Behaviour Therapy (CBT) especially designed for fatigued cancer patients is an effective treatment.

Aim: To identify and measure (neuro)physiological factors of fatigue in fatigued cancer survivors and to determine the role of these factors in the maintaining of fatigue. The identification of (neuro)physiological factors of persistent fatigue can help to improve the diagnostics of fatigue, predict therapy outcome and facilitate other treatment options. Finally, if (neuro)physiological characteristics of fatigue can be influenced by CBT it will enhance our understanding of the mechanism causing fatigue.

Research questions: 1) What are characteristic (neuro)physiological factors of fatigue in disease-free cancer patients? 2) To which degree can these factors be influenced by Cognitive Behaviour Therapy?

Design: In this explorative study fatigued disease-free cancer patients (n=57), who finished treatment for cancer at least one year and maximally ten years ago, will be approached for this study and asked for informed consent. They will be compared to age and sex matched non-fatigued patients (n=21). First, a base-line assessment will take place, which includes magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) to assess brain morphology and brain metabolites, respectively. To assess peripheral and central fatigue a two-minute endurance test will be administered at maximal voluntary (isometric) contraction (MVC). During the test changes in EMG and force indicate peripheral fatigue, while central fatigue is studied by the twitch interpolation technique. A maximal exercise test will be performed to assess physical fitness and deconditioning. At baseline patients will also be given an actometer which will register daily activity during two weeks. Further, the actometer will register daily activity up to five days after the maximal exercise test. Finally, at baseline patients will fill out a standardized questionnaire, including the Checklist Individual Strength and a self-observation list to assess fatigue severity. Then, the fatigued patients start immediately with Cognitive Behaviour Therapy (CBT). At the end of the therapy, after 6 months, a second assessment will take place in this group of patients. The assessment consists of the same measurements as at baseline. The results will be compared with the baseline situation to analyze the effect of CBT on the (neuro)physiological parameters.

Relevance of this study: Fatigue long after treatment for cancer is a frequently occurring problem, which has important consequences for quality of life in these patients. Identification of characteristic (neuro)physiological factors of fatigue in disease-free cancer patients may not only serve a theoretical understanding of this invalidating condition, but may also provide an objective biological marker that could support the diagnosis and follow-up of treatment. The identification of (neuro)physiological factors which play a role in fatigue after cancer may aid in the early recognition of patients who are at risk for developing fatigue and may lead to early intervention and/or different treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Treated for a malignant solid tumour.
* Completion of treatment for cancer minimal 1 year ago
* Single treatment modality surgery permitted
* Current hormonal therapy permitted
* Disease-free, as defined by the absence of somatic disease activity parameters.
* Age between 19 and 65.
* Age at disease onset minimal 18 years

Exclusion Criteria:

* Brain tumour in the past
* Current psychological or psychiatric treatment.
* Physical comorbidity which could explain the fatigue.
* Contra-indication for MR examinations (e.g. claustrophobia).
* Treatment with anti-depressive drugs, anti-epileptic drugs, benzodiazepines.
* Insufficient command of the Dutch language to fill out questionnaires.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Possible (neuro)physiological determinants of postcancer fatigue | The measurements will be performed at baseline and comparable measurements will be performed 6 months later (after 6 months cognitive behavior therapy or 6 months waiting list condition)
  MRI to assess brain morphology; MRS to assess brain metabolite concentrations; sEMG and force registration to assess central and peripheral muscle fatigue; maximal exercise test to assess physical condition; actometer measurements and self-observation list to assess daily activity and symptoms; standardized questionnaires to assess fatigue severity and general health; neurological tests to assess information processing and motor speed; screening of blood and urine to find possible explanations for postcancer fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: H.W.M. van Laarhoven, Md, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Derived] Muller F, Wijayanto F, Abrahams H, Gielissen M, Prinsen H, Braamse A, van Laarhoven HWM, Groot P, Heskes T, Knoop H. Potential mechanisms of the fatigue-reducing effect of cognitive-behavioral therapy in cancer survivors: Three randomized controlled trials. Psychooncology. 2021 Sep;30(9):1476-1484. doi: 10.1002/pon.5710. Epub 2021 May 3. PMID 33899978
- [Derived] Ter Veer E, Prinsen H, Sprangers MAG, Zwinderman KAH, Bleijenberg G, van der Pouw Kraan TCTM, de Vries IJM, Wierenga EA, van Laarhoven HWM. Interferon Gamma-Induced Protein (IP-10) as Potential Biomarker for Cancer-Related-Fatigue: Results from a 6-month Randomized Controlled Trial. Cancer Invest. 2018;36(7):371-377. doi: 10.1080/07357907.2018.1499933. Epub 2018 Sep 6. PMID 30188739
- [Derived] Prinsen H, Heerschap A, Bleijenberg G, Zwarts MJ, Leer JW, van Asten JJ, van der Graaf M, Rijpkema M, van Laarhoven HW. Magnetic resonance spectroscopic imaging and volumetric measurements of the brain in patients with postcancer fatigue: a randomized controlled trial. PLoS One. 2013 Sep 11;8(9):e74638. doi: 10.1371/journal.pone.0074638. eCollection 2013. PMID 24040301
- [Derived] Prinsen H, Bleijenberg G, Heijmen L, Zwarts MJ, Leer JW, Heerschap A, Hopman MT, van Laarhoven HW. The role of physical activity and physical fitness in postcancer fatigue: a randomized controlled trial. Support Care Cancer. 2013 Aug;21(8):2279-88. doi: 10.1007/s00520-013-1784-9. Epub 2013 Mar 22. PMID 23519566
- [Derived] Prinsen H, Bleijenberg G, Zwarts MJ, Hopman MT, Heerschap A, van Laarhoven HW. Physiological and neurophysiological determinants of postcancer fatigue: design of a randomized controlled trial. BMC Cancer. 2012 Jun 18;12:256. doi: 10.1186/1471-2407-12-256. PMID 22708881